CLINICAL TRIAL: NCT01031914
Title: Evaluation of an Algorithm to Detect Sleep and Wake in Continuous Positive Airway Pressure Users Using Paced Breathing
Brief Title: Evaluation of an Algorithm to Detect Sleep and Wake in Continuous Positive Airway Pressure (CPAP)
Acronym: PBSW
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Philips Respironics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: AR-0931-PBSW-SS
Record Dates: First submitted 2009-12-11; First posted 2009-12-15 (Estimated); Results first posted 2013-05-14 (Estimated); Last update posted 2013-05-14 (Estimated); Status verified 2013-04

CONDITIONS: Sleep Apnea, Obstructive
Keywords: Paced Breathing; OSA; sleep/wake detection
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Paced Breathing Sleep/Wake detection (Experimental): All subjects enrolled will have oobstructive sleep apnea (OSA) and will be current Continuous Positive Airway Pressur (CPAP) users.
  Interventions: Device: Paced Breathing

INTERVENTIONS:
Device: Paced Breathing — The Paced Breathing (PB) feature(when activated) will work to relax the user and help them fall asleep by encouraging them to take deep slow breaths until they reach 10 breaths (or less) per minute. The feature will also detect when the subject has fallen asleep so the Continuous Positive Airway Pressur (CPAP) device will automatically switch from PB mode to regular CPAP mode.
  Other Names: Respironics

SUMMARY:
The purpose of this engineering trial is to develop and validate an algorithm that will deliver Paced Breathing as a ramp feature to obstructive sleep apnea (OSA) subjects using Continuous Positive Airway Pressure (CPAP) therapy. In this trial the investigators will be evaluating the algorithm's ability to correctly distinguish between sleep and wake.

ELIGIBILITY:
Inclusion Criteria:

* Age 21-70
* Diagnosis of obstructive sleep apnea (OSA)
* Current adherent CPAP user (has been using CPAP nightly for at least 2 weeks).
* On CPAP pressures of 5-10cm.
* Subjects wishing to complete a day or evening appointment need to have significant daytime sleepiness (Epworth Sleepiness Scale score of 8 or above)
* Able and willing to provide written informed consent
* English speaking

Exclusion Criteria:

* Participation in another interventional research study within the last 30 days
* Major controlled or uncontrolled medical condition such as congestive heart failure, neuromuscular disease, renal failure etc.
* Inability to tolerate nasal CPAP mask due to problems breathing solely through their nose.
* Chronic respiratory failure or insufficiency with suspected or known neuromuscular disease, moderate or severe chronic obstructive pulmonary disease (COPD), or any condition with an elevation of arterial carbon dioxide levels while awake (PaCo2≥55mmHg)
* Severe oxygen desaturation on the polysomnography (PSG), i.e. Sa02 < 70% for 10% of the study.
* Surgery of the upper airway, nose, sinus or middle ear within the past 90 days
* Currently using supplemental oxygen
* Regular use of sleeping pills or stimulants (> 3 nights a week)
* Currently working night shift or rotating day/night shift
* Drowsy Driving or near miss accident in the past 6 months
* Inability to tolerate or track to Paced Breathing device during initial habituation session in lab
* Chronic insomnia, Restless legs syndrome, or severe periodic limb movement disorder (PLMD - PLMAI>20/hr).

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2009-10; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David P White, M.D, Principal Investigator — Philips Respironics
Locations (1):
- Philips Respironics, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from the general population, the sleep clinic at Sleep HealthCenters, Only subjects who had a diagnostic polysomnography and who were CPAP for at least 2 weeks, were considered for inclusion. Informed consent were be obtained by an investigator or research coordinator and was required for enrollment into the study.
Pre-assignment Details: N/A All participants enrolled in the trial have completed the study
Groups:
- Paced Breathing Sleep/Wake Detection: All subjects enrolled will have obstructive sleep apnea (OSA) and will be current CPAP users.
Period: Overall Study
Arm/Group | Paced Breathing Sleep/Wake Detection
Started | 36
Completed | 36
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Paced Breathing Sleep/Wake Detection: All subjects enrolled will have OSA and will be current CPAP users.
Arm/Group | Paced Breathing Sleep/Wake Detection
Number analyzed (Participants) | 36
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 35
  >=65 years | 1
Age Continuous [Mean (Standard Deviation); unit: years] | 48.1 (11.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 25
Region of Enrollment [Number; unit: participants]
  United States | 36

OUTCOME MEASURES:

1. Primary Outcome: Sleep/Wake Algorithm
Description: We tested the ability of the Sleep/Wake algorithm to identify sleep an wake periods with precision, as compared to standard polysonography (PSG) measures, which was used as the gold standard, i.e. we tested the accuracy of the algorithm. Accuracy was defined as the proportion of true results (both true positives and true negatives)in the population and it was assesed using as 2 X 2 table, i.e. accuracy = number of true positives + number of true negatives/ number of true positives + false positives + false negatives +true negatives. where True positive = the algorithm tested correctly identified sleep, False positive = the algorithm tested incorrectly identified sleep, True negative = the algorithm tested correctly rejected awake periods, and False negative = the algorithm tested incorrectly rejected awake periods.
Time Frame: The performance of the algorithm will be evaluated in real time while the subject is wearing the device during the sleep study, an average of 08 hours.
Population: All the participants completing the sleep study were included in the analysis
Measure: Number; unit: accuracy (%)
Arm/Group | Paced Breathing Sleep/Wake Detection
Number analyzed (Participants) | 36
accuracy (%) | 62

ADVERSE EVENTS:
Time Frame: Adverse events were recorded through the duration of the sleep study, an average of 8 hours.
Arm/Group | Paced Breathing Sleep/Wake Detection
Serious Adverse Events (participants affected / at risk) | 0/36
Other Adverse Events (participants affected / at risk) | 10/36
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Paced Breathing Sleep/Wake Detection (N=36)
Central Sleep apnea (Nervous system disorders) | 10 (10)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes